CLINICAL TRIAL: NCT05616780
Title: Does Severity of Airflow Obstruction Correlate to Static Lung Volumes Obtained by Nitrogen Washout and Body Plethysmography?
Brief Title: Does Severity of Airflow Obstruction Correlate to Static Lung Volumes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Hawkins (Other)
Responsible Party: Sponsor-Investigator, Virginia Hawkins, Chief Investigator, Manchester Metropolitan University
Organization: Manchester Metropolitan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 46246
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: airflow obstruction, plethysmography, lung volumes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obtaining lung volume measurements in patients with airflow obstruction (Other): All patients involved in this study will be attending a pulmonary function test as part of their routine patient treatment pathway, requested by their consultant. Potential participants will be sent a patient information sheet prior to their lung function test.
  The pulmonary function test begins routinely, with the pre-test questions. Spirometry will then be performed. If the patient's results are variable and the repeatability criteria are not met, the patient will not be asked to take part in the study, and no additional tests (not requested by the consultant routinely) will be carried out. If the patient has normal or obstructive results (FEV1/FVC <70%) the patient will sign the consent form and both lung volume tests will be conducted. They must be able to follow the instructions for both nitrogen washout and body plethysmography, and the results must also meet the acceptability and repeatability criteria.
  Interventions: Other: Physiological test

INTERVENTIONS:
Other: Physiological test — Lung volume measurements will be obtained using nitrogen washout and body plethysmography

SUMMARY:
Obstructive lung disease is defined by limitations in expiratory airflow, caused by excess mucus, loss of muscle tone, and structural changes. Over time airflow reduction can lead to gas trapping in the lungs (hyperinflation). Hyperinflation is linked to diminished exercise tolerance, shortness of breath, and a poor quality of life. Early treatment options include inhalers and pulmonary rehabilitation; however, surgical intervention and oxygen therapy may be required in the later stages. More prompt, accurate diagnosis will help to improve patient outcomes and optimise their treatment pathways.

Two methodologies used to determine lung volumes and hyperinflation, are nitrogen washout and body plethysmography. The accuracy of each in defining lung volumes in patients with obstructive lung disease is debated in literature. Plethysmography requires the patient to sit in an enclosed box and perform a panting manoeuvre and uses measured changes in volume and pressure to derive lung volumes. Plethysmography has been suggested to overestimate lung volumes in patients with obstructive lung disease. On the other hand, nitrogen washout relies on 'washing out' all the nitrogen from the lungs to calculate lung volumes. Gas trapping and poor airflow circulation that occurs in patients with airflow obstruction may lead to underestimated lung volumes.

This study will aim to investigate if there is a significant difference between lung volumes obtained by both nitrogen washout and body plethysmography in patients with obstructive lung disease. Subjects with mild, moderate, severe, and very severe obstruction, including those with no obstruction for comparison will be included, with approximately 10 from each group. They will be asked if they consent to undergo an extra test during their routine hospital appointment, which will add ~15 minutes to their visit.

DETAILED DESCRIPTION:
Obstructive lung disease is defined by limitations in expiratory airflow, caused by excess mucus, loss of muscle tone, and structural changes. Over time airflow reduction can lead to gas trapping in the lungs (hyperinflation). Hyperinflation is linked to diminished exercise tolerance, shortness of breath, and a poor quality of life. Early treatment options include inhalers and pulmonary rehabilitation; however, surgical intervention and oxygen therapy may be required in the later stages. More prompt, accurate diagnosis will help to improve patient outcomes and optimise their treatment pathways.

Two methodologies used to determine lung volumes and hyperinflation, are nitrogen washout and body plethysmography. The accuracy of each in defining lung volumes in patients with obstructive lung disease is debated in literature. Plethysmography requires the patient to sit in an enclosed box and perform a panting manoeuvre and uses measured changes in volume and pressure to derive lung volumes. Plethysmography has been suggested to overestimate lung volumes in patients with obstructive lung disease. On the other hand, nitrogen washout relies on 'washing out' all the nitrogen from the lungs to calculate lung volumes. Gas trapping and poor airflow circulation that occurs in patients with airflow obstruction may lead to underestimated lung volumes.

This study will aim to investigate if there is a significant difference between lung volumes obtained by both nitrogen washout and body plethysmography in patients with obstructive lung disease. Subjects with mild, moderate, severe, and very severe obstruction, including those with no obstruction for comparison will be included, with approximately 10 from each group. They will be asked if they consent to undergo an extra test during their routine hospital appointment, which will add ~15 minutes to their visit.

Expiratory airflow limitation is the hallmark of obstructive pulmonary disease; Parenchymal remodelling, mucous impaction, oedema, and a decrease of smooth muscle tone all contribute to the structural and anatomical changes that occur (O'Donnell, 2006). Individuals with bronchiectasis and chronic obstructive pulmonary disease often have inflammation in their airways (COPD). Impaired mucociliary clearance and increased mucus production are caused by inflammation that occurs inside the airway epithelium. Because of increased connective tissue deposition, the bronchial walls thicken, and the lumen of the airways decrease over time (Hogg, 2004). Airflow obstruction is defined as a reduction in expiratory airflow when compared to the total volume of air exhaled and is investigated by a test called spirometry. The two measurements required to identify obstructive lung disease are FEV1 (forced expiratory volume in the first second of expiration following a maximal inspiration) and FVC (forced vital capacity - the maximal amount of air that can be exhaled forcibly following maximal inhalation). For airflow obstruction to be diagnosed the FEV1/FVC ratio of must be <70%. The FEV1 percent predicted is then used to determine the severity of obstruction following this. Spirometry is commonly used to identify the presence of COPD (chronic obstruction pulmonary disease) or the severity/absence of obstruction in diseases such as asthma (Eschenbacher, 2016). TLC (total lung capacity) describes the amount of air in the lungs at maximal inspiration, the expected amount is determined by height, age, weight, ethnicity and gender. Chest wall deformities, tumours, level of physical activity and the presence of respiratory disease can all alter an individual's TLC.

Often, as a result of chronic obstructive lung disease, hyperinflation occurs which is the abnormal increase in FRC. This is caused by the imbalance between the reduction in airflow from the lungs compared to the total volume of the lungs. Changes in elastic properties of the lungs and impaired inspiratory muscle function also contribute to the extent of hyperinflation over time (Gibson, 1996). Hyperinflation is associated with reduced exercise capacity, dyspnoea and reduced quality of life. Individuals with COPD were found to spend 1/3 of the day standing/walking compared to healthy individuals of the same age who spent around ½ of the day doing so; such physical deconditioning significantly accelerates disease progression (Cooper, 2009). Treatment and intervention that targets hyperinflation can improve not only respiratory symptoms but also metabolic parameters and chronic inflammation. Pulmonary rehabilitation, bronchodilators and oxygen therapy are often utilised, however, surgical intervention such as lung volume reduction surgery (LVRS) is believed to provide the most benefit (Criner, 2017). The accuracy of lung volume measurements is vital to determine if interventional treatment (e.g., bronchodilators, LVRS, supplemental oxygen) have been successful or if a patient needs surgical intervention.

Methods including body plethysmography, nitrogen washout, helium dilution, and the more novel radiographic method utilising computed tomography (CT) are used by clinicians to calculate lung volumes. They produce measurements comprising FRC (functional residual capacity), IC (inspiratory capacity), and VC (vital capacity) which are used to calculate TLC (Delgado, 2019). Figure 1 gives a schematic of how these values relate to each other. The two methods that are investigated in this research project are nitrogen washout and body plethysmography. Nitrogen washout is a gas dilution technique that involves the patient breathing 100% oxygen through a mouthpiece to remove the nitrogen from the lungs. The mouthpiece has a two-way valve allowing the patient to breathe in oxygen whilst exhale through a pneumotach that measures the concentration of nitrogen in the exhaled air until it reaches <1.5% (Wanger, 2005). Body plethysmography measures pressure variations in a chamber with a constant temperature and volume. The patient must perform several breathing manoeuvres, including tidal breathing and panting, through a pneumotach inside an air-tight chamber. Chest wall collapse and expansion alters the pressure within the chamber, this is measured by transducers and allows lung volume measurements to be taken (Delgado, 2019).

There has long been debate over the accuracy of lung volume measurement techniques, Garfield et al stated that body plethysmography overestimates lung volumes in patients with airway obstruction in comparison to CT (Garfield, 2012). Lufti et al more recently stated in their research gas dilution techniques like nitrogen washout may underestimate TLC in patients with obstructive lung disease (Lutfi, 2017). One case study looking at lung volumes in a single patient with obstructive lung disease suggested that plethysmography may falsely elevate lung volume measurements due to airway resistance and mouth compliance, whereas nitrogen washout might underestimate volumes due to non-communicative areas of the lungs (Sue, 2013). On the other hand, another study found, when comparing lung volumes derived from CT to body plethysmography and helium dilution, in patients with obstructive lung disease, there was a significant difference between CT and helium dilution but not CT and body plethysmography (O'Donnell CR, 2010), suggesting plethysmography was the more accurate of the two. As helium dilution and nitrogen washout both rely on gases mixing to determine lung volumes, perhaps similar results may be seen if this was repeated using nitrogen washout. To the researcher's knowledge there has not been a comparison between lung volumes obtained via nitrogen washout and body plethysmography in patients with varying severities of obstructive lung disease. If a significant difference is found between the methods, this could aid in choosing the most appropriate and accurate lung volume measurement tool in patients with obstructive lung disease. Such findings may shorten appointment times, improve patient treatment pathways and reduce monetary costs to the hospital. COPD costs the NHS approximately 1.9 billion a year, earlier intervention and treatment may help to reduce this burden (The_Lancet, 2018).

ELIGIBILITY:
Inclusion Criteria:

A minimum of 10 patients from each group will be included; normal lung function/ no airflow obstruction (FEV1/FVC >70%), mild airflow obstruction (FEV1/FVC <70% and FEV1 >80% predicted), moderate airflow obstruction (FEV1/FVC <70% and FEV1 50-80% predicted), severe airflow obstruction (FEV1/FVC <70% and FEV1 30-50% predicted) and very severe (FEV1/FVC <70% and FEV1 >30% predicted).

Al patients will be over the age of 18 with no upper age limit. No children will be included in this study.

Patients must have withheld their inhalers.

Exclusion Criteria:

[15:10] Jessica Armstrong

Contraindications to performing the test include (if occurred within last 8 weeks):

* Heart attack
* Stroke
* Haemoptysis
* Pneumothorax
* Surgery to the abdomen/thorax
* Eye surgery

An individuals spirometry cannot be included if:

* There is a cough during the first second of the manoeuvre
* A leak at the mouthpiece
* Early termination of manoeuvre
* Sub optimal effort
* They are unable to comprehend the instructions
* Obstruction of the mouthpiece (tongue/teeth)

Lung volume measurements cannot be included if:

* There is a leak around the mouthpiece
* The patient has a ruptured eardrum
* They are unable to comprehend the instructions
* Obstruction of the mouthpiece (tongue/teeth)
* The patient is on supplementary oxygen and cannot come off it (this must be discontinued for a suitable period prior to nitrogen washout)
* Patients who are CO2 retainers may not be able to undergo nitrogen washout

The patients test results must meet the acceptability criteria of the ARTP pulmonary function testing statement (updated 2020). For spirometry this states that there must be 3 technically acceptable attempts within 150ml, however, if the the individual has an FVC <1.00L this can be 100ml. Nitrogen washout requires two technically acceptable attempts within 10% (as per trust policy), whereas, for body plethysmography three technically acceptable attempts should be obtained within 5%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Measurement of lung volumes by two routine techniques in patients referred for pulmonary function testing. | 6 months
  Patients referred for pulmonary function test as part of their routine patient treatment pathway will have lung volumes measured by nitrogen washout and body plethysmography, which are both routine techniques. Participants will have a range of obstructive or normal lung function. When the test is finished, patients will be told that their test results will be sent to their consultant, who will then explain them at a follow up appointment/ phone call (this is routine procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas John, Principal Investigator — Shrewsbury and Telford Hospital Trust
Locations (1):
- Shrewsbury and Telford hospital Trust, Telford, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No